CLINICAL TRIAL: NCT06295679
Title: A Real-world, Prospective, Observational Study Assessing the Effectiveness of Repatha® Used in Combination With Standard of Care Compared With Standard of Care Alone on Major Cardiovascular Events in Chinese Patients With Established Atherosclerotic Cardiovascular Disease
Brief Title: A Study Assessing Repatha® in Combination With Standard of Care (SOC) Compared With SOC on Major Cardiovascular Events in Chinese Participants With Atherosclerotic Cardiovascular Disease
Status: Recruiting | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20180442
Record Dates: First submitted 2024-02-26; First posted 2024-03-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Major Cardiovascular Event; Established Atherosclerotic Cardiovascular Disease
Keywords: Cardiovascular death; Myocardial infarction; Stroke; Unstable angina; Coronary revascularization; Atherosclerotic Cardiovascular Disease; Repatha
MeSH Terms: conditions — Myocardial Infarction; Stroke; Angina, Unstable; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Repatha® with Standard of Care Exposure: Participants with clinically evident ASCVD treated with Repatha® in combination with SOC in a clinical setting. To ensure that the recruitment strategy has as little impact on routine practice as possible, the decision to treat the participant with Repatha® with SOC will be made independently of, and before, enrollment in the study.
- Standard of Care Exposure: Participants with clinically evident ASCVD treated with SOC alone in a clinical setting. To ensure that the recruitment strategy has as little impact on routine practice as possible, the decision to treat the participant with SOC only will be made independently of, and before, enrollment in the study.

SUMMARY:
The primary objective of the study is to evaluate real-world effectiveness of treatment with Repatha® in combination with SOC, compared with SOC alone, on the risk for cardiovascular (CV) death, myocardial infarction (MI), stroke, hospitalization for unstable angina, or coronary revascularization, whichever occurs first, in participants with established atherosclerotic CV disease (ASCVD) treated with SOC, according to local clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants ≥ 18 years of age.
* Participants or participant's legally authorized representative has provided informed consent to participate in this study.
* Participants who meet one of the following:
* Prescribed Repatha® in addition to an existing SOC treatment according to local guidelines and approved label.

OR

* Already received SOC treatment prior to enrollment.
* Participants with ANY of the following.
* Diagnosis of MI OR stroke within 2 years before enrollment.
* 2 MIs OR ≥ 2 strokes OR (≥ 1 MI AND ≥ 1 stroke) any time before enrollment.
* Diagnosis of (MI OR stroke) AND diabetes.
* Diagnosis of (MI OR stroke) AND documented multivessel disease (defined as > 50% stenosis of ≥ 2 major coronary arteries on coronary angiography or coronary artery contrast enhanced computed tomography).
* Diagnosis of symptomatic peripheral arterial disease.
* Most recent fasting LDL-C ≥ 70 mg/dL (≥ 1.8 mmol/L) or nonhigh-density lipoprotein cholesterol (non-HDL-C) ≥ 100 mg/dL (≥ 2.6 mmol/L) within 6 months prior to enrollment.
* Most recent fasting triglycerides ≤ 400 mg/dL (≤ 4.5 mmol/L) within 6 months prior to enrollment.

Exclusion Criteria:

* Stroke within past 1 month.
* Known hemorrhagic stroke at any time.
* Stroke due to thromboembolic event.
* Any prior use of Repatha® or other proprotein convertase subtilisin/kexin type 9 inhibition treatments within past 6 months prior to enrollment.
* Participants currently enrolled in another study involving any investigational procedure, device or drug.
* Participants prescribed Repatha® with a history of severe hypersensitivity or allergy to any subsidiary.

Ages: 18 Years to 150 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises Chinese participants with established ASCVD treated with Repatha® in combination with SOC or with SOC alone in a clinical setting which includes any primary through tertiary healthcare setting where Repatha® is prescribed.
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2022-12-19 (Actual); Primary Completion 2028-12-19 (Estimated); Study Completion 2028-12-19 (Estimated)

PRIMARY OUTCOMES:
Time to CV Death, MI, Hospitalization for Unstable Angina, Stroke, or Coronary Revascularization, Whichever Occurs First | Up to 72 months

SECONDARY OUTCOMES:
Time to CV Death, MI, or Stroke, Whichever Occurs First | Up to 72 months
Change in Low-density Lipoprotein Cholesterol (LDL-C) From Baseline | Baseline and end of follow-up (up to 72 months)
Percent Change in LDL-C From Baseline | Baseline and end of follow-up (up to 72 months)
Number of Participants Who Experienced Adverse Events | Up to 72 months
Number of Participants Who Experienced Adverse Drug Reactions | Up to 72 months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (89):
- China (89):
  - China Japan Friendship Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Fuwai Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Haidian Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Chongqing Emergency Medical Center, Chongqing, Chongqing Municipality
  - Chongqing General Hospital, Chongqing, Chongqing Municipality
  - Dongguan Songshan Lake Central Hospital, Dongguan, Guangdong
  - The First Peoples Hospital of Foshan, Foshan, Guangdong
  - The First Affiliated Hospital Sun-Yat Sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Shantou University Medical College, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Nanfang Hospital Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital Sun Yat-sen University, Guangzhou, Guangdong
  - The Third Peoples Hospital of Huizhou, Huizhou, Guangdong
  - Zhuhai Peoples Hospital, Zhuhai, Guangdong
  - The Second Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - The First Peoples Hospital of Yulin, Yulin, Guangxi
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Tangshan Gongren Hospital, Tangshan, Hebei
  - Heilongjiang Provincial Hospital, Haerbin, Heilongjiang
  - The Fourth Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Huaihe Hospital of Henan University, Kaifeng, Henan
  - Nanyang Central Hospital, Nanyang, Henan
  - The Seventh Peoples Hospital of Zhengzhou, Zhengzhou, Henan
  - Fuwai Central China Cardiovascular Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Central Hospital of Wuhan, Wuhan, Hubei
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Wuhan No 1 Hospital, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical college, Huazhong University of Science and Technology, Wuhan, Hubei
  - Wuhan Third Hospital-Tongren Hospital of Wuhan University, Wuhan, Hubei
  - Hunan Provincial Peoples Hospital, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Changshu No1 Peoples Hospital, Changshu, Jiangsu
  - Changshu No2 Peoples Hospital, Changshu, Jiangsu
  - Nantong First Peoples Hospital, Nantong, Jiangsu
  - The First Peoples Hospital of Kunshan, Suzhou, Jiangsu
  - Wuxi Peoples Hospital, Wuxi, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Jiangxi Provincial Peoples Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Nanchang, Nanchang, Jiangxi
  - The Second Norman Bethune Hospital of Jilin University, Changchun, Jilin
  - Central Hospital of Dalian University of Technology (Dalian Municipal Central Hospital), Dalian, Liaoning
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - General Hospital of Northern Theater Command, Shenyang, Liaoning
  - The Fourth Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Tangdu Hospital of Air Force Medical University, Xi'an, Shaanxi
  - Shaanxi Provincial Peoples Hospital, Xi'an, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Jinan Central Hospital, Jinan, Shandong
  - The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong
  - Provincial Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - Affiliated hospital of Jining Medical University, Jining, Shandong
  - Zibo central Hospital, Zibo, Shandong
  - Tongji Hospital of Tongji University, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated To Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi An Jiaotong University, Xi’an, Shanxi
  - Sichuan Academy of Medical Sciences Sichuan Provincial Peoples Hospital, Chengdu, Sichuan
  - Chengdu First Peoples Hospital, Chengdu, Sichuan
  - Chengdu Third Peoples Hospital, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin Peoples Hospital, Tianjin, Tianjin Municipality
  - Tianjin First Central Hospital, Tianjin, Tianjin Municipality
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Yanan Hospital of Kunming City, Kunming, Yunnan
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First Peoples Hospital of Yunnan Province, Kunming, Yunnan
  - Sir Run Run Shaw Hospital Affiliated to Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - the First Peoples Hospital of Xiaoshan District Hangzhou, Hangzhou, Zhejiang
  - Huzhou Central Hospital, Huzhou, Zhejiang
  - The First Peoples Hospital of Huzhou, Huzhou, Zhejiang
  - Jiaxing Second Hospital, Jiaxing, Zhejiang
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang
  - Shaoxing Second Hospital, Shaoxing, Zhejiang
  - Beijing Anzhen Hospital, Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com